CLINICAL TRIAL: NCT01777373
Title: Conducting Airways in Lung Fibrosis
Brief Title: Conducting Airways in Lung Fibrosis (VACFI)
Acronym: VACFI
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P110902; N° IDRCB : 2012-A00295-38 (Other: AFSSAPS)
Record Dates: First submitted 2012-10-02; First posted 2013-01-28 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2014-12

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: conducting airway, bronchiolization
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Idiopathic pulmonary fibrosis (IPF): Idiopathic pulmonary fibrosis (IPF)
- Control: Control
- Non-IPF interstitial lung disease (ILD): Non-IPF interstitial lung disease (ILD)
- Uncharacterized ILD: Uncharacterized ILD

SUMMARY:
The purpose of this study is to determine whether extension of the conducting airways into the distal lung, or bronchiolization, occurs early in the course of Idiopathic Pulmonary Fibrosis, a disease wherein normal lung structures are destroyed and replaced by non-functional scar tissue.

DETAILED DESCRIPTION:
Diffuse Interstitial Pneumonias are a heterogeneous group of chronic respiratory diseases. Idiopathic Pulmonary Fibrosis, one of such diseases, is characterized by lesions of the conducting airways including extension of bronchioles towards the distal lung, or bronchiolization of the distal lung. Such lesions are traditionally referred to as "traction bronchiectasis" although no evidence supports a cause-and-effect relationship between alveolar fibrosis and airway lesions. Another feature of IPF is chronic, invalidating dry cough. Our hypothesis is that IPF is characterized by early increases in the volume of conducting airways, that such changes correlate with cough, and that airway changes are in direct relation with airway fibrosis. The primary aim of this study is to demonstrate increased anatomical dead space (VD), a surrogate for conducting airway volume, in patients with moderate (or early) IPF, in comparison with subjects without any respiratory disease ("non-DIP controls"). The secondary aims are : To show that VD is increased in patients with IPF in comparison with patients with other DIPs ("DIP controls"), to show that in patients with IPF increased VD does not correlate with indices of alveolar fibrosis, and to show associations between increased VD and cough and other respiratory symptoms in patients with IPF.

ELIGIBILITY:
IPF :

INCLUSION CRITERIA

1. Age 18-85 years
2. IPF diagnosed according to ATS/ERS/JRS/ALAT criteria
3. Patient gave informed consent

NON INCLUSION CRITERIA

1. Presence of respiratory comorbidities : Asthma, COPD, bronchiectasis, emphysema, tuberculosis sequelae, prior lung surgery
2. Obstructive ventilatory disorder
3. Counterindication to pulmonary function testing
4. Women : Pregnancy or milking
5. Lack of health insurance

Controls :

INCLUSION CRITERIA

1. Volunteers aged 18-85 years, free of any respiratory disease
2. Volunteer gave informed consent

Secondary EXCLUSION CRITERIA Abnormal PFT : Total lung capacity or FEV1/VC ratio < Lower Limit of Normal

Non-IPF ILD :

INCLUSION CRITERIA

1. Age 18-85 years
2. Radiological interstitial pneumonia, on 2 tests performed >3 months apart
3. PINS histology OR sarcoidosis histology OR clinical diagnosis of drug-induced lung disease OR diagnosis of auto-immune disease
4. Patient gave informed consent

NON INCLUSION CRITERIA

1. Presence of respiratory comorbidities : Asthma, COPD, bronchiectasis, emphysema, tuberculosis sequelae, prior lung surgery
2. Obstructive ventilatory disorder
3. Counterindication to pulmonary function testing
4. Women : Pregnancy or milking
5. Lack of health insurance

Uncharacterized ILD :

INCLUSION CRITERIA

1. Age 18-85 years
2. Radiological interstitial pneumonia, on 2 tests performed >3 months apart
3. Patient gave informed consent

NON INCLUSION CRITERIA

1. Presence of respiratory comorbidities : Asthma, COPD, bronchiectasis, emphysema, tuberculosis sequelae, prior lung surgery
2. Obstructive ventilatory disorder
3. Counterindication to pulmonary function testing
4. Women : Pregnancy or milking
5. Lack of health insurance

Secondary EXCLUSION CRITERIA Final diagnosis other than either IPF or non-IPF interstitial pneumonia.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: IPF will be diagnosed according to ATS/ERS/JRS/ALAT 2012 guidelines, either in the presence of a typical Usual Interstitial Pneumonia pattern on CT imaging of the lung or in the presence of a probable UIP pattern on a pathological lung specimen, and in the absence of any identified cause of secondary interstitial pneumonia.
  Patients with non-IPF interstitial pneumonias will be recruited. Due to the case mix at Bichat and Pompidou hospitals, patients with idiopathic Non Specific Interstitial Pneumonia and interstitial pneumonia associated with sarcoidosis and auto-immune disease will be recruited.
  In some patients, a definitive diagnosis of either IPF or non-IPF interstitial pneumonia will not be available at the time of inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2012-08; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Fowler dead space | 1 day
  Conducting airway volume is determined by Fowler's method from volumetric capnography data

SECONDARY OUTCOMES:
Bohr anatomic dead space | 1 day
  Bohr anatomic dead space is determined from capnography and spirometry data.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent PLANTIER, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Bichat, Paris, France